CLINICAL TRIAL: NCT00202813
Title: The Use of Antibiotic-coated Venous Catheters in the Critically Ill Child: Reducing the Rate of Bloodstream Related Infections
Brief Title: Study of the Use of Coated Venous Catheters in the Critically Ill Child
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corewell Health West (Other)
Collaborators: Helen DeVos Children's Hospital (Other)
Responsible Party: Principal Investigator, Robert Fitzgerald, Pediatric Critical Care Physician, Corewell Health West
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2003-104
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Children in the Pediatric Intensive Care Unit or General Pediatric Care Unit Requiring a Central Venous Catheter
Keywords: CVC; central venous catheter; infection; bloodstream infection; catheter infection; pediatric; children; antibiotic impregnated catheters
MeSH Terms: conditions — Infections; Sepsis

INTERVENTIONS:
Device: Cook Spectrum Pediatric Central Venous Catheter Anti-microbial Impregnated Polyurethane and Arrow Pediatric Central Venous Catheter

SUMMARY:
This study should help determine to determine whether or not the use of an antibiotic coated catheter will significantly reduce the number of central line related bloodstream infections in children requiring a CVC. This study may also determine if antibiotic coated catheters will be significantly less likely than non-antibiotic coated catheters to allow bacteria to live (colonize) in/on the catheter.

The use of central venous catheters (CVC) is paramount to the care of critically ill children. Thus, in the pediatric intensive care unit (PICU), these catheters are widely used in situations when more than peripheral venous access is necessary. This central access allows the delivery of fluids, e.g, blood, medications, etc. as well as serves as a means to withdraw blood. It has been estimated that more than 250,000 nosocomial bloodstream infections occur each year, with 90% of these associated with the use of CVCs. More recently, the National Nosocomial Infection Surveillance System (NNIS) reported during 1992-2001 CVC-associated bloodstream infections (BSI) in ICU settings occurred at rates of 2.9-11.3 BSI per 1,000 catheter days. The cost of treating CVC related BSI has been estimated to be in excess of $28,000 per catheter. In the adult medical literature, there is strong evidence supporting use of antiseptic or antibiotic coated catheters to reduce the cost of hospitalization for CVC related infections. Cost-benefit studies have suggested that if the baseline incidence of CVC BSI is >0.4 BSI per 1000 catheter days, $59,000 will be saved, 7 cases of BSI will be avoided, and 1 death prevented for every 300 anti-septic impregnated CVCs used.

DETAILED DESCRIPTION:
Catheter related infections are often difficult to treat because the pathogen may form a biofilm that actually embeds itself into the catheter material. Additionally, the catheter hub and skin around this area may be colonized with bacteria. It is by this route that pathogenic organisms migrate to the external surface of the catheter, which then can progress to the intravascular tip. To decrease the risk of CVC associated infections, antibiotic coated catheters have been used. Since 1990, several types of antiseptic or antimicrobial vascular catheters have been developed. These catheters are designed to protect both the external and internal surfaces of the device from colonization of certain bacteria. Raad et al, have demonstrated in a randomized multicenter clinical trial among hospitalized adult patients that CVCs coated with minocycline and rifampin significantly reduced the risk for catheter-related colonization and bloodstream infections[8]. However, there have been no clinical trials reported in the pediatric population on this issue. This study will prospectively compare in a randomized, blinded fashion the use of two Food & Drug Administration (FDA) approved central venous catheters - an antibiotic coated CVC to non-coated CVC at DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan. Additional major pediatric teaching hospitals may be added at a later time.

ELIGIBILITY:
Inclusion Criteria:

all patients ages 21 years or less admitted to the pediatric intensive care unit or general pediatric unit at DeVos Children's Hospital

research informed consent must be signed

Exclusion Criteria:

known allergy or sensitivity to minocycline, tetracyline, doxycycline, oxytetracycline, demeclocycline, rifampin, rifabutin

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500
Dates: Start 2003-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
to determine if antibiotic coated catheters reduce the risk of catheter associated BSI in children hospitalized in PICU or in inpatient pediatric ward in comparison to non-antibiotic coated catheters.
An infection free interval is defined as beginning with the insertion of the cvc (or, if applicable with the cure of a infection in a catheter that was left in place anbd concluded with one of the outcomes listed

SECONDARY OUTCOMES:
to determine the bacterial pathogens associated with antibiotic coated CVC BSI and compare these pathogens with those normally associated with non-antibiotic coated CVC
To determine the bacterial pathogens associated with colonization of antibiotic coated catheter tips in comparison to those normally associated with non-antibiotic coated catheter tips.
To determine risk factors associated with CVC BSI

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fitzgerald, MD, Principal Investigator — Helen DeVos Children's Hospital
Locations (1):
- DeVos Children's Hospital, Grand Rapids, Michigan, United States